CLINICAL TRIAL: NCT05102279
Title: Analysis of Urine Composition Saturation and Dietary Intervention in Subjects Without Urinary Calculi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Ding Feng, professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UUC-2021-10
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Calculi, Urinary; Dietary Supplements; Urine Specimen Collection
Keywords: Dietary Supplements; Urine Saturation factor; Calculi, Urinary
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Intervention Model Description: Participants were randomly divided into two groups.A group of participants first received a normal phosphorus diet for 2 days, followed by a low-phosphorus diet for 3 days, then a normal phosphorus diet for 2 days, and a high-phosphorus diet for 3 days.The other group of participants first received a normal phosphorus diet for 2 days, followed by a high phosphorus diet for 3 days, then a normal phosphorus diet for 2 days, and a low phosphorus diet for 3 days.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early administration of high-phosphorus diet test group (Experimental): Group A: 1500 mg phosphorus diet was given on day 1-2, 2500 mg phosphorus diet on day 3-5, 1500 mg phosphorus diet on day 6-7 and 500 mg phosphorus diet on day 8-10
  Interventions: Dietary Supplement: Giving subjects different phosphorus diets at different stages of the trial
- Early administration of low-phosphorus diet test group (Active Comparator): Group B: 1500 mg phosphorus diet was given on day 1-2, 500 mg phosphorus diet on day 3-5, 1500 mg phosphorus diet on day 6-7 and 3500 mg phosphorus diet on day 8-10
  Interventions: Dietary Supplement: Giving subjects different phosphorus diets at different stages of the trial

INTERVENTIONS:
Dietary Supplement: Giving subjects different phosphorus diets at different stages of the trial — Ordinary phosphorus diet: Phosphorus content 1500mg High phosphorus diet: Phosphorus content 2500mg (inorganic phosphorus is added to the ordinary phosphorus diet) Low phosphorus diet: Phosphorus content 500mg (Protein content is achieved through chicken albumen and addition of low-phosphorus whey protein powder) The ratio of plant protein and animal protein is the same as the other two diets. In addition, calcium-magnesium tablets and potassium chloride salt are added to achieve the same calcium, magnesium and potassium content as the other two diets.) There are 2 recipes for each diet. Ensure that the energy, protein, fat, carbohydrate, calcium, magnesium, sodium, potassium, oxalic acid content, vegetable protein and animal protein ratio are basically the same: Energy: 2100kcal (30kcal/kg, standard body weight 70kg) Protein: 110g Fat: 55-60g Carbohydrate: 300g Calcium: 600-700mg Magnesium: 350-400mg Sodium: 4600mg Potassium: 2500mg

SUMMARY:
Urinary calculi have become a global public health problem, which brings a huge economic burden to society and individuals. The pathogenesis of urinary calculi is not completely clear. Supersaturation of urinary components is a necessary condition for the formation of urinary calculi. The causes of stone formation are closely related to diet, drugs, metabolic disorders, basic diseases, genetic factors, environment and so on. Diet essentially determines the composition of urine, which affects the formation of urinary calculi. The effect of dietary phosphorus intake on stones is not clear. There is a lack of data to support dietary phosphorus as an influencing factor of stone formation. Phosphorus is present in most foods. 24h urine composition analysis is of great value in predicting the occurrence and composition of urinary calculi. However, due to the interaction between urine components, a single urine component can not well predict the occurrence of stones. Therefore, the researchers introduced the relative supersaturation of common stone components in urine to predict the incidence of stones. Therefore, we want to give healthy adults a diet with different phosphorus content for a period of time to clarify the effect of phosphorus in the diet on 24h urine composition level and urine relative supersaturation, so as to further explore the relationship between dietary phosphorus and the incidence of urinary calculi. To provide more clear recommendations for early prevention of urinary calculi, and provide more evidence for clinical decision-making, thereby reducing the incidence rate of urinary calculi.

DETAILED DESCRIPTION:
*Diet: Ordinary phosphorus diet: phosphorus content 1500mg High-phosphorus diet: Phosphorus content is 2500mg (inorganic phosphorus is added to the ordinary phosphorus diet) Low-phosphorus diet: Phosphorus content 500mg (The protein content and the ratio of plant protein and animal protein are consistent with the other two diets by adding egg protein and adding low-phosphorus whey protein powder. In addition, calcium magnesium tablets and potassium chloride salt are added to achieve the same calcium, magnesium and potassium content as others. The two diets are consistent)

There are 2 recipes for each diet, and each recipe guarantees that the energy, protein, fat, carbohydrate, calcium, magnesium, sodium, potassium, oxalic acid content, vegetable protein and animal protein ratio are basically the same:

Energy: 2100kcal (30kcal/kg, standard weight 70kg);Protein: 110g;Fat: 55-60g;Carbohydrate: 300g;Calcium: 600-700mg;Magnesium: 350-400mg;Sodium: 4600mg;Potassium: 2500mg Water:Giving subjects 2L of purified water without any minerals every day

* Specimen We will collect 24h urine and feces for the whole day on the 2nd, 5th, 7th, and 10th days of the experiment, and collected morning blood and random urine on the 3rd, 6th, 8th, and 11th days.
* Analysis We will use Equil 2 software to calculate the relative supersaturation of urine, and use SPSS software to analysis data

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-45 years old
* 18. 5≤Body Mass Index≤ 23. 9
* Normal oral diet

Exclusion Criteria:

* People who have had or are suffering from urinary tract stones , or have the following diseases leading to the formation of stones: renal tubular acidosis, gout, hyperuricemia, chronic diarrhea, insulin resistance, hyperparathyroidism, idiopathic hypercalcemia, hypertension, diabetes mellitus
* CKD-EPI-eGFR<90ml/min1.73m-2)
* The following drugs are being used: cathartic, aspirin, angiotensin converting enzyme inhibitor，angiotensin II receptor antagonist，diuretic, acid inhibitor, alkali or carbonic anhydrase inhibitor, phosphorus binder, calcium agent and active vitamin D;
* Previous gastrointestinal diseases or gastrointestinal surgery
* Application of enteral and parenteral nutrition
* Complicated with infection, with or without antibiotic treatment
* Mental patients or unable to cooperate for various reasons

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Subjects complete the trial within 10 days | 10 days
  Subjects ate all the food during the trial period and collected all specimens

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ding, PhD, Study Director — Division of Nephrology,Shanghai Ninth People's Hospital
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635
- [Background] Shadman A, Bastani B. Kidney Calculi: Pathophysiology and as a Systemic Disorder. Iran J Kidney Dis. 2017 May;11(3):180-191. PMID 28575878
- [Background] Prezioso D, Strazzullo P, Lotti T, Bianchi G, Borghi L, Caione P, Carini M, Caudarella R, Ferraro M, Gambaro G, Gelosa M, Guttilla A, Illiano E, Martino M, Meschi T, Messa P, Miano R, Napodano G, Nouvenne A, Rendina D, Rocco F, Rosa M, Sanseverino R, Salerno A, Spatafora S, Tasca A, Ticinesi A, Travaglini F, Trinchieri A, Vespasiani G, Zattoni F; CLU Working Group. Dietary treatment of urinary risk factors for renal stone formation. A review of CLU Working Group. Arch Ital Urol Androl. 2015 Jul 7;87(2):105-20. doi: 10.4081/aiua.2015.2.105. PMID 26150027
- [Background] Peacock M. Phosphate Metabolism in Health and Disease. Calcif Tissue Int. 2021 Jan;108(1):3-15. doi: 10.1007/s00223-020-00686-3. Epub 2020 Apr 7. PMID 32266417